CLINICAL TRIAL: NCT02381080
Title: A Drug-drug Interaction Study of Ibrutinib With Moderate and Strong CYP3A Inhibitors in Patients With B-cell Malignancy
Brief Title: Interaction Study of Ibrutinib and Cytochrome P450 (CYP) 3A Inhibitors in Participants With B-cell Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR106609; PCI-32765LYM1003 (Other: Janssen Research & Development, LLC); 2015-000325-36 (EudraCT Number)
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
Keywords: B-Cell Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma; Waldenstrom's Macroglobulinemia; Ibrutinib; IMBRUVICA; PCI-32765; JNJ-54179060
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Waldenstrom Macroglobulinemia | interventions — ibrutinib; Erythromycin; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Part 1: Ibrutinib+Erythromycin+Voriconazole (Experimental): Participants will receive oral treatment in six, 28-days cycles. In Cycle 1, participants will take ibrutinib 560 milligram (mg) (4*140 mg capsules) once daily (QD) from Days 1- 4; on Days 5-11 ibrutinib 140 mg capsule QD in combination with erythromycin 500 mg tablet 3 times daily (TID); on Days 12-13 ibrutinib 140 mg capsule QD; on Days 14-18 ibrutinib 560 mg (4*140 mg capsules) QD; on Days 19-25 ibrutinib 140 mg capsule QD in combination with voriconazole 200 mg tablet twice daily (BD); on Days 26-27 ibrutinib 140 mg capsule orally QD; and on Day 28 and in subsequent treatment Cycles (2-6) participants will continue oral treatment with ibrutinib 420 mg or 560 mg QD (depending on the subtype of B-cell malignancy).
  Interventions: Drug: Ibrutinib; Drug: Erythromycin; Drug: Voriconazole
- Part 2: Ibrutinib+ Erythromycin+Voriconazole (Experimental): Participants will receive oral treatment in six, 28-days cycles. In Cycle 1, participants will take ibrutinib 560 mg (4*140 mg capsules) QD from Days 1- 4; on Days 5-18 ibrutinib 560 mg (4*140 mg capsules) QD in combination with either erythromycin 500 mg tablet TID (Group 1) or voriconazole 200 mg tablet BD (Group 2); on Day 19 and in subsequent treatment Cycles (2-6) participants will continue oral treatment with ibrutinib 420 mg or 560 mg QD (depending on the subtype of B-cell malignancy).
  Interventions: Drug: Ibrutinib; Drug: Erythromycin; Drug: Voriconazole

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib capsule (at dose level of 140 or 420 or 560 mg) will be taken orally QD up to six, 28-days cycles.
  Other Names: Imbruvica; PCI-32765; JNJ-54179060
Drug: Erythromycin — Erythromycin 500 mg tablet will be taken orally TID (Part1 Cycle 1: on Days 5-10 and morning dose on Day 11; Part2 Cycle 1: on Days 5-17 and morning dose on Day 18).
  Other Names: Erythrocin
Drug: Voriconazole — Voriconazole 200 mg tablet will be taken orally BD (Part1 Cycle 1: on Days 19-25; Part2 Cycle 1: on Days 5-17).
  Other Names: VFEND

SUMMARY:
The purpose of this study is to assess the effect of a moderate Cytochrome P450 (CYP) 3A inhibitor (erythromycin) and a strong CYP3A inhibitor (voriconazole) on the steady-state pharmacokinetics (PK [the study of the way a drug enters and leaves the blood and tissues over time]) of repeated oral doses of ibrutinib in participants with B-cell malignancy (cancer or other progressively enlarging and spreading tumors).

DETAILED DESCRIPTION:
This is an open-label (participants and researchers are aware about the treatment participants are receiving), multi-center (when more than 1 hospital or medical school team work on a medical research study), drug-drug interaction (DDI) study of ibrutinib with the moderate and the strong CYP3A inhibitors (erythromycin and voriconazole respectively) in participants with B-cell malignancies (including Chronic Lymphocytic Leukemia /Small Lymphocytic Lymphoma [CLL/SLL], Follicular Lymphoma [FL], Marginal Zone Lymphoma [MZL], Waldenstrom's Macroglobulinemia [WM] or Mantle Cell Lymphoma [MCL]). The study will consist of a Screening Phase (28 days), a Treatment Phase (consisting of six 28-days cycles), and an End-of-Treatment (EoT) Visit (within 30 days after the last dose of study drug). The study will consist of 2 Parts. In Part 1, extent of the DDI between ibrutinib at dose level of 140 milligram (mg) and CYP3A inhibitors will be assessed. After completion of Part 1 of the study, an interim analysis of all available PK and safety data will be conducted and Part 2 will only be performed if the observed drug interaction is less than anticipated based on current information. In Part 2, safety and PK of ibrutinib at dose level of 560 mg administered with CYP3A inhibitors will be assessed. Participants who continue to derive clinical benefit from ibrutinib treatment at the end of this study, and who are eligible to continue in the PCI-32765CAN3001 study (NCT01804686) will end their participation in this trial, have an EoT visit completed, and will continue receiving ibrutinib as a part of the PCI-32765CAN3001 protocol. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Chronic Lymphocytic Leukemia /Small Lymphocytic Lymphoma (CLL/SLL), Marginal Zone Lymphoma (MZL), Mantle Cell Lymphoma (MCL), Follicular Lymphoma (FL), or Waldenstrom's Macroglobulinemia (WM)
* Relapsed or refractory disease after at least 1 prior line of systemic therapy (participants with FL or MZL must have failed anti-CD20 monoclonal antibody containing chemotherapy regimen)
* Eastern Cooperative Oncology Group Performance Status score of 0 or 1
* Hematology values within the following limits: a) Absolute neutrophil count (ANC) greater than and equal to (>=) 1.0*10^9 per liter (L); b) Platelets >=50*10^9/L without transfusion support within 7 days; c) Hemoglobin >=8 gram per deciliter (g/dL) without transfusion support within 7 days; d) Prothrombin time /International normalized ratio (PT/INR) less than equal to (<=) 1.5*Upper Limit of Normal (ULN) and activated partial thromboplastin time (aPTT) <=1.5*ULN
* Biochemical values within the following limits: a) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <=3.0*ULN; b) Total bilirubin <=1.5*ULN (unless due to Gilbert's syndrome); c) Serum creatinine <=1.5*ULN or a calculated creatinine clearance of >=50 milliliter per minute per 1.73 square meter

Exclusion Criteria:

* Major surgery within 4 weeks of the first dose of ibrutinib
* Diagnosed or treated for malignancy other than the indication under study except for: a) Adequately treated non-melanoma skin cancer or lentigo maligna, curatively treated in-situ cancer without evidence of disease; b) Malignancy treated with curative intent and with no known active disease present for >=3 years before the first dose of ibrutinib
* History of stroke or intracranial hemorrhage within 6 months prior to the first dose of ibrutinib
* History of galactose intolerance
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists (for example, phenprocoumon)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-05-19 (Actual); Primary Completion 2016-06-24 (Actual); Study Completion 2016-06-24 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Ibrutinib | Cycle 1: 0 hour (hr) pre-dose on Day 1; 0 hr pre-dose, 0.5,1,2,3,4,6,8 and 24 hrs post-dose on Day 4, 11, 18, and 25
  The Cmax is the maximum observed plasma concentration.
Minimum Observed Plasma Concentration (Cmin) of Ibrutinib | Cycle 1: 0 hour (hr) pre-dose on Day 1; 0 hr pre-dose, 0.5,1,2,3,4,6,8 and 24 hrs post-dose on Day 4, 11, 18, and 25
  The Cmin is the minimum observed plasma concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Ibrutinib | Cycle 1: 0 hour (hr) pre-dose on Day 1; 0 hr pre-dose, 0.5,1,2,3,4,6,8 and 24 hrs post-dose on Day 4, 11, 18, and 25
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC[0-24]) of Ibrutinib | Cycle 1: 0 hr pre-dose, 0.5,1,2,3,4,6,8 and 24 hrs post-dose on Day 4, 11, 18, and 25
  The AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours.
Metabolite to Parent (M/P) Ratio of Ibrutinib | Cycle 1: 0 hour (hr) pre-dose on Day 1; 0 hr pre-dose, 0.5,1,2,3,4,6,8 and 24 hrs post-dose on Day 4, 11, 18, and 25
  Ratio of ibrutinib metabolite concentration to parent compound (ibrutinib) concentration will be assessed.

SECONDARY OUTCOMES:
Partial Area Under the Plasma Concentration-Time Curve Between 2 Defined Timepoints (AUC [t1 and t2]) of Voriconazole | Cycle 1: 0 hour (hr) pre-dose on Day 5; 0 hr pre-dose, 0.5,1,2,3,4,6 and 24 hrs post-dose on Day 18 and 25
  The AUC (t1 and t2) is the partial area under the plasma concentration-time curve from time 't1' to 't2' hours.
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening up to end of study (up to 8 months)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. An SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trials, Study Director — Janssen Research & Development, LLC
Locations (6):
- N/a N/a, Canada
- Russia (3):
  - Moscow
  - Petrozavodsk
  - Saint Petersburg
- Spain (2):
  - Madrid
  - Pamplona

REFERENCES:
- See also: A Drug-Drug Interaction Study of Ibrutinib With Moderate and Strong CYP3A Inhibitors in Patients With B-cell Malignancy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=9493&filename=CR106609_CSR.pdf